CLINICAL TRIAL: NCT01220076
Title: Phase II Study Evaluating According to the Polymorphism of CYP2D6, the Rate of Biological Response to Treatment With Tamoxifen (TAM) Administered in Pre-operative Situation in Patients With Breast Cancer Non Metastatic HR+
Brief Title: Biological Response to Tamoxifen (TAM) in Patients With Breast Cancer Non Metastatic RH+
Acronym: TAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BRD 08/11-A
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Non Metastatic Breast Cancer
Keywords: Tamoxifen,; Breat Cancer; Pharmacogenetic; non metastatic breast cancer, HR +
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tamoxifene (Experimental)
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: tamoxifen

SUMMARY:
The biological response to treatment with tamoxifen in the preoperative situation is studying in this protocol. This study will enrolls patients with non-metastatic breast cancer HR +.

The relationship between the CYP2D6 polymorphism, pharmacokinetics and biological efficacy of TAM will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult Females (≥ 18 years), with effective contraception. The contraceptive should not use estrogen to a derivative. It must be continued during treatment with tamoxifen for at least two months after his arrest.
* Histologically confirmed diagnosis of invasive breast cancer, previously untreated. Patients have been supported for a breast cancer may be included if a period of at least 2 years between the last systemic treatment of inclusion in the study.
* Primary tumor hormonopositive: ER and / or PR ≥ 50% by immunohistochemistry.
* Lack of HER2 overexpression
* Palpable primary tumor or greater than or equal to 20 mm in diameter, measured by ultrasound
* Patient scheduled to undergo breast cancer surgery
* No metastases
* Clinical Stage M0
* Performance index ≤ 1 (OMS)
* Neutrophils WBC > or = 1500 / mm3, Platelets > or = 100 000/mm3 Hemoglobin ≥10 g/dL
* Normal liver function: bilirubin ≤ 1.5 x ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases).
* Normal renal function (creatinine ≤ 1.5 mg / dL or creatinine clearance ≥ 60 mL / min)
* Cardiac function (MUGA scan or ultrasound February> 55%) and lung function, 5.2.2 Criteria related to participation in the study:
* Patient affiliated to social security, Patient has signed and dated consent

Non-Inclusion Criteria:

1. Pregnant or Breastfeeding women
2. Use of St. John's Wort (herbal tea ...) within 5 days before starting treatment
3. Consumption of grapefruit juice in the last 5 days of starting treatment
4. Congenital galactosemia
5. Glucose and galactose malabsorption
6. Lactase deficiency
7. Co-medications that may interfere with cytochrome P450:
8. Ongoing Enzyme inducers:

   * Antiepileptic drugs: carbamazepine, phenobarbital, phenytoin
   * Antinfectieux: rifampin, rifabutin, névrirapine, griséofilvine, efavirenz
9. Ongoing Enzyme Inhibitors:

   * Inhibitors of serotonin reuptake: fluoxetine, paroxetine
   * Thioridazine. Quinidine
   * Amiodarone
   * Ca antagonists: diltiazem, verapamil
   * azole antifungals ketoconazole, fluconazole, miconazole.
   * No protease inhibitors: ritonavir, nelfinavir, amprenavir, indinavir.
   * Macrolides: erythromycin, clarithromycin, josamycin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the response to Tamoxifen treatment, in preoperative situations (immediately operable patients) in patients with positive Hormone Receptors (HR+) non-metastatic breast cancer | 5 weeks
  The primary endpoint is the determination of the variation in the KI-67 expression, a marker of cell proliferation, at the tumour level between the initial biopsy (T0) and after 5 weeks of tamoxifen treatment, in relation to cytochrome 2D6 polymorphisms. A 50% geometric reduction in KI-67 expression at 5 to 7 weeks should be considered as a major response

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Léon Berard, Lyon
  - Institut Curie, Paris
  - Institut de Cancerologie de l'Ouest (ICO), Saint-Herblain